CLINICAL TRIAL: NCT03146026
Title: The Effects of a 12- Week Combined Exercise Training Program on Arterial Stiffness, Endothelial Function, Inflammatory Markers and Metabolic Profile in Obese Adolescent Girls: A Pilot Study.
Brief Title: The Effects of a Combined Exercise Training Program on Vascular Health and Metabolic Profile in Obese Adolescent Girls.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PusanNU-2
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Obesity, Adolescent
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Exercise (CON) (No Intervention): Fifteen obese adolescent girls. This arm did not perform any exercise training for 12 weeks. Caloric intake was 1921.7 kcal/day.
- Combined Exercise Training (CET) (Experimental): Fifteen obese adolescent girls. This arm performed combined exercise training 3 times per a week for 12 weeks. Caloric intake was 1921.7 kcal/day.
  Interventions: Behavioral: Combined Exercise Training

INTERVENTIONS:
Behavioral: Combined Exercise Training — The CET program was performed for 60 minutes with 5 minutes of warm-up and cool-down per day, 3 times a week for 12 weeks. Combined exercise consisted of 20 minutes of various resistant band exercises (Upper body: seated rows, biceps curl, shoulder flexion, elbow flexion, chest press; Lower body: hip flexion, hip extension, calf raise, leg press, squat) and 30 minutes of treadmill walking. The warm-up and cool down consisted of static stretching. Intensity of exercise was gradually increased from 40-50% heart rate reserve (HRR) in weeks 1-4, and to 60-70% HRR in weeks 9-12. Each training session was fully supervised by the researchers. Every subject wore a heart rate monitor during the whole training session so as to maintain the correct training intensity.
  Arms: Combined Exercise Training (CET)

SUMMARY:
The purpose of this study was to examine the impact of 12 weeks of combined exercise training (CET) on arterial stiffness, endothelial function, inflammatory markers, insulin resistance, and body composition in obese adolescent girls. Thirty obese adolescent girls participated in this study. The girls were randomly divided into CET group (n=15) and control group (n=15). The CET group performed concurrent resistance training followed by aerobic training at 40-70% of the heart rate reserves (HRR) 3 days/week for 12 weeks. Plasma nitric oxide, endothelin-1, C-reactive protein, arterial stiffness, homeostasis model assessment of insulin resistance (HOMA-IR), glucose, insulin, and the adiponectin/leptin ratio were measured before and after the 12-weeks study.

ELIGIBILITY:
Inclusion Criteria:

* Obese with hyperinsulinemia
* Abdominal obesity
* Sedentary (no regular exercise training or physical activity)
* No weight loss diet during last 6 months.

Exclusion Criteria:

* Hypertension
* Pregnancy
* Chronic disease

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2011-05-02 (Actual); Study Completion 2011-05-06 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | 12 weeks
  Arterial stiffness was measured as measurement of baPWV (m/s).
Endothelin-1 | 12 weeks
  Levels of Endothelin-1 in blood were measured by Endothelin-1 enzyme immunoassay kit.
Insulin resistance | 12 weeks
  Insulin resistance was estimated using the homeostasis model assessment of insulin resistance (HOMA-IR).
Plasma leptin | 12 weeks
  Plasma leptin was determined by ELISA kit
Plasma adiponectin | 12 weeks
  Plasma adiponectin was measured using ELISA kit
Body weight | 12 weeks
  Body weight was measured to nearest 0.1 kg.
Height | 12 weeks
  Height was measured to nearest 1 cm.
Waist circumference | 12 weeks
  Waist circumference was measured at midpoint between the lower rib and the iliac crest at the end of a normal expiration using a tape measure
Body fat | 12 weeks
  Percent body fat (%) was determined using a bioelectrical impedance-meter.
Maximal heart rate | 12 weeks
  Maximal heart rate was obtained at the end of a graded treadmill exercise test performed until volitional exhaustion.
Nitric oxide | 12 weeks
  Nitric oxide generation was measured by Griess assay kit.

REFERENCES:
- [Derived] Wong A, Sanchez-Gonzalez MA, Son WM, Kwak YS, Park SY. The Effects of a 12-Week Combined Exercise Training Program on Arterial Stiffness, Vasoactive Substances, Inflammatory Markers, Metabolic Profile, and Body Composition in Obese Adolescent Girls. Pediatr Exerc Sci. 2018 Nov 1;30(4):480-486. doi: 10.1123/pes.2017-0198. Epub 2018 Sep 7. PMID 30193554